CLINICAL TRIAL: NCT00583193
Title: A Study of the Effectiveness and Tolerability of Duloxetine (Cymbalta) in the Treatment of PTSD.
Brief Title: Open-Label Duloxetine Monotherapy in the Treatment of Posttraumatic Stress Disorder
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Canive, Jose M., M.D. (Individual)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Jose M. Canive, M.D., New Mexico VA Health Care System
Organization: New Mexico VA Healthcare System (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F1J-US-X024
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2007-12-31 (Estimated); Status verified 2007-12

CONDITIONS: Posttraumatic Stress Disorders
Keywords: Post Traumatic Stress Disorder; Duloxetine; Antidepressants
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Open-label Study
  Interventions: Drug: Duloxetine hydrochloride

INTERVENTIONS:
Drug: Duloxetine hydrochloride — Start 30 mg Q.D. for 7 days, then increased to 60 mg Q.D. @ the week 1 visit. Thereafter, dose may be increased or decreased by 30 mg increments based on tolerability and efficacy between a dosage range of 60 to 120 mg.
  Other Names: Cymbalta

SUMMARY:
The purpose of this study is to determine whether Duloxetine (Cymbalta®) is an effective treatment in reducing the symptoms of Posttraumatic Stress Disorder (PTSD).

DETAILED DESCRIPTION:
Duloxetine has established efficacy for treatment of major depression, generalized anxiety disorder and diabetic peripheral neuropathic pain. Chronic PTSD is often treated with antidepressants, in fact there are only two FDA-approved treatments for PTSD. Yet many chronic PTSD patients, especially male combat veterans, have a limited response to antidepressant treatment (Baker et al, 1995; Cañive et al, 1998; Hertzsberg et al 2000) and new pharmacotherapies should be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ages 18 or older of any ethnic background meeting DSM-IV criteria for PTSD
* Score of at least 60 on the CAPS-SX at baseline
* Competent to give informed consent
* If female, patient should be using a medically approved contraceptive, or not otherwise be of childbearing potential
* Patients who have not taken medications or herbal remedies for a psychiatric indication within one week prior to the baseline visit (treatment phase); two weeks prior in the case of fluoxetine or in the case of an MAOI
* Other medications, if any, must have been kept stable for at least one month prior to the baseline visit

Exclusion Criteria:

* Known hypersensitivity to duloxetine or any of the inactive ingredients
* Females who are pregnant or breastfeeding
* Use of antipsychotics, antidepressants, or benzodiazepines (except for short-term use during study as specified in Concomitant Medications section) within one week prior to the baseline visit and throughout the study period
* Use of fluoxetine or an MAOI within two weeks
* Concomitant use of narrow therapeutic index medications or medications that are likely to have a clinically significant drug interaction with duloxetine
* Medical conditions that may prevent safe administration of duloxetine including end stage renal disease, clinically significant renal impairment (CrCl <30 mL/min), hepatic insufficiency, cardiac disease, or pulmonary disease
* Patients with uncontrolled narrow-angle glaucoma
* Alcohol or drug abuse or dependence within three months of study entry as defined by DSM-IV criteria
* Alcohol use may not exceed 12 drinks per week or 5 drinks per drinking episode during the course of the study.
* A current or past history of bipolar disorder, schizophrenia, schizoaffective disorder or other psychotic disorder
* Suicidal or homicidal ideation or other clinically significant dangerous behavior
* Currently seeking compensation or increase in compensation for the effects of the trauma
* Initiation or change in psychotherapy within 3 months of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-12; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
PTSD Symptoms will be assessed by the Clinician-Administered PTSD Scale for DSM-IV (CAPS) | Performed at baseline, weeks 1, 2, 4, 8, & 12

SECONDARY OUTCOMES:
Visual Analog Scale for Pain (VAS) | Baseline, weeks 1, 2, 4, 8, & 12

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Canive, M.D., Principal Investigator — New Mexico VA Healthcare System
Locations (1):
- New Mexico VA Health Care System, Albuquerque, New Mexico, United States